CLINICAL TRIAL: NCT05835635
Title: Level of Satisfaction and Quality of Life in People Living With HIV in Chile, Who Switch From Oral Therapy to Long-acting Injectable Cabotegravir + Rilpivirine
Brief Title: Switch From Oral Therapy to Long-acting Injectable Cabotegravir + Rilpivirine
Acronym: CABO-LA
Status: Not yet recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Maria Elena Ceballos, MD, Assistant Professor School of Medicine, Pontificia Universidad Catolica de Chile
Other Study IDs: 220817002
Record Dates: First submitted 2023-03-24; First posted 2023-04-28 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Patient Satisfaction; Patient Preference; Quality of Life; Acceptability of Health Care
Keywords: Quality of life; Acceptability; Satisfaction; Preference; HIV; Long acting- cabotegravir
MeSH Terms: conditions — Patient Satisfaction; Patient Preference; Patient Acceptance of Health Care; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol will assess the level of satisfaction, acceptance of treatment and quality of life of patients with undetectable HIV who voluntarily change from oral to injectable antiretroviral treatment at 72 weeks of follow-up.

DETAILED DESCRIPTION:
Foreign studies have shown that long-acting (LA) injectable Cabotegravir + Rilpivirine is effective and well tolerated in the long term, demonstrating non-inferiority in relation to oral antiretroviral therapy. One of the main advantages described is that patients report a better quality of life and greater satisfaction with their new antiretroviral therapy.

Currently in Chile, HIV patients have only access to oral antiretroviral therapy as part of their health coverage, either in public ( FONASA) or at private ( ISAPRES). Several issues regarding oral antiretroviral therapy have been detected, including: a) patients who have been in treatment for a long time, often complain of being tired of taking 1 or more pills daily, which might directly affect adherence and success of treatment, b) some patients complain about gastrointestinal intolerance, associated with oral therapy; and c) patients who have to travel abroad for longer than a month, have problems to get an extra dose, in order to adhere to their antiretroviral treatment.

That is why, the possibility of receiving a bimonthly injectable antiretroviral therapy, becomes an attractive alternative for our patients.

Studies evaluating efficacy and security of LA-injectable Cabotegravir + rilpivirine were ATLAS, ATLAS-2M and FLAIR. ATLAS and ATLAS-2M only included 26 and 45 Latin American patients (Argentina and Mexico) from a total of 616 and 1045 participants, respectively. FLAIR study did not include Latin American individuals. Since the majority of patients included in the registration studies were not of Hispanic or Latino ethnicities, it is important to evaluate, in population living in Chile, the real-life impact of Cabotegravir + Rilpivirine injectable treatment on the level of satisfaction, in experienced patients and how it will affect them in the long-term period.

Injectable therapy with Cabotegravir + Rilpivirine needs to be administered by a third person, in an authorized place for such procedures, and requires refrigeration. For this reason, starting the program as a part of a study facilitates the logistic implementation of such program.

The objective of this study is to evaluate, in real life, the level of satisfaction, acceptance of treatment, and quality of life in a group of HIV patients treated in HIV consultation at Red Salud UC-Christus, in Santiago de Chile, who switch to LA injectable therapy Cabotegravir + Rilpivirine, during a 72 weeks follow-up. In order to measure these items, the investigators will use validated instruments (questionnaires).

III. Hypotheses The change from oral to injectable antiretroviral therapy in HIV patients is associated with a high level of satisfaction, good acceptance of treatment, and better quality of life, without affecting adherence to treatment, keeping undetectable HIV viral load an stable CD4 count, and with few serious adverse effects related to injectable therapy.

IV. Objectives Primary Objective: Evaluate the level of satisfaction, acceptance of treatment, and quality of life of undetectable HIV patients who switch from oral to injectable antiretroviral treatment at 72 weeks follow up

Secondary Objectives:

1. Describe percentage of patients that preferred injectable over oral therapy after 72 weeks follow up
2. Evaluate the adherence of patients switching to injectable treatment
3. Evaluate safety/tolerability of the injectable treatment
4. Monitor the HIV viral load, of the patients every 6 months, to follow their health status
5. Monitor the CD4 count of the patients every 6 months, to follow their health status 6 Monitor blood chemistry of the patients every 6 months, to follow their health status

7. Register anthropometric changes.

ELIGIBILITY:
Inclusion Criteria:

All patients who, according to the recommendations for use, can receive LA- injectable Cabotegravir +Rilpivirine therapy will be invited to participate in the study.

Recommendations for use:

* HIV-1 positive patients, on antiretroviral therapy
* Older than 18 years of age at the time of signing the informed consent
* Undetectable HIV viral load in the last 6 months
* Willing to switch from oral to injectable therapy

Exclusion Criteria:

These criteria are defined for those patients who, according to the recommendations for use, cannot receive the therapy:

* Previous virological failure
* Any evidence of primary resistance or the presence of any major known INI or NNRTI resistance-associated mutation by any historical resistance test result.
* Patients with decompensated pathology (physical or mental) or active opportunistic infection at the time of admission
* Concomitant use with: rifampin, carbamazepine, oxcarbazepine, phenytoin and phenobarbital or any contraindication to one of the drugs of the study
* Known hepatitis B co-infection
* Pregnancy (There is insufficient data for people who become pregnant on CAB or those planning to conceive because available pregnancy PK data are limited (n = 3), and data on clinical outcomes in pregnancy are extremely limited. Therefore, CAB is Not Recommended for pregnant or nonpregnant people initiating or restarting ART or for those whose current regimen is not well tolerated and/or not fully suppressive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV patients who meet the inclusion criteria and who are willing to switch from oral to injectable therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the level of satisfaction of undetectable HIV patients who switch from oral to injectable antiretroviral treatment at 72 weeks follow up. | 72 weeks
  Level of satisfaction of HIV treatment will be measured by HIVTSQs (HIV Treatment Satisfaction Questionnaire) at day one, week 4,12, 36,52 and 72. Questionnaire produce a Treatment Satisfaction score (range: 0 to 66). The higher the score, the greater the satisfaction with treatment.
Evaluate the level of acceptance of treatment of undetectable HIV patients who switch from oral to injectable antiretroviral treatment at 72 weeks follow up. | 72 weeks
  Acceptance of treatment will be measured by ACCEPT questionnaire (Chronic Treatment Acceptance Questionnaire) at day 1, week 36 and week 72. Questionnaire score has ranges from 0 to 66. The higher the score, indicates greater acceptance
Evaluate the level of quality of life of undetectable HIV patients who switch from oral to injectable antiretroviral treatment at 72 weeks follow up. | 72 weeks
  Quality of life will be evaluated by MOS-HIV (Medical Outcomes Study HIV Health Survey) Questionnaires at day 1, weeks 4,36,60 and 72. Questionnaire score has ranges from 0 to 100. The higher the score, indicates better health

SECONDARY OUTCOMES:
Evaluate the adherence of patients switching to injectable treatment | 72 weeks
  Patient adherence will be measured at 72 weeks, through the number of injections that the patient attends.
Evaluate safety of the injectable treatment | From day 28 to 72 weeks
  The evaluation of safety will be monitored through incidence of All Drug related AEs and SAEs, AEs leading to discontinuations
Describe percentage of patients who prefer injectable over oral therapy at 72 weeks follow up | 72 weeks
  Patient´s preference will be described by "SOLAR preference questionnaire" at week 72 by the percentaqe of patients that prefer injectable over oral therapy
Monitor the HIV viral load of the patients every 6 months, to follow their health status | Every 6 months until 72 weeks
  HIV-1 RNA by Copies RNA/mL will be registrered at day 1, week 20, 52, and 72.
Monitor the lymphocytes CD4 count of the patients every 6 months, to follow their health status | Every 6 months until 72 weeks
  Absolute Values for lymphocytes CD4 Count by cells/mm3 will be registered at day 1, week 20, 52, and 72.
Monitor the blood chemistry of the patients every 6 months, to follow their health status | Every 6 months until 72 weeks
  Blood chemistry includes creatinine, SGOT, GGT, SGPT, alkaline phosphatases and bilirrubin at day 1, week 20, 52, and 72.
Register anthropometric changes | From day 1 to 72 weeks
  Height, weight and hip measures will be registered at day 1, week 20, 52, and 72.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Ceballos, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- CICUC, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Result] Scarsi KK, Swindells S. The Promise of Improved Adherence With Long-Acting Antiretroviral Therapy: What Are the Data? J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:23259582211009011. doi: 10.1177/23259582211009011. PMID 33902356
- [Result] Swindells S, Andrade-Villanueva JF, Richmond GJ, Rizzardini G, Baumgarten A, Masia M, Latiff G, Pokrovsky V, Bredeek F, Smith G, Cahn P, Kim YS, Ford SL, Talarico CL, Patel P, Chounta V, Crauwels H, Parys W, Vanveggel S, Mrus J, Huang J, Harrington CM, Hudson KJ, Margolis DA, Smith KY, Williams PE, Spreen WR. Long-Acting Cabotegravir and Rilpivirine for Maintenance of HIV-1 Suppression. N Engl J Med. 2020 Mar 19;382(12):1112-1123. doi: 10.1056/NEJMoa1904398. Epub 2020 Mar 4. PMID 32130809
- [Result] Overton ET, Richmond G, Rizzardini G, Jaeger H, Orrell C, Nagimova F, Bredeek F, Garcia Deltoro M, Swindells S, Andrade-Villanueva JF, Wong A, Khuong-Josses MA, Van Solingen-Ristea R, van Eygen V, Crauwels H, Ford S, Talarico C, Benn P, Wang Y, Hudson KJ, Chounta V, Cutrell A, Patel P, Shaefer M, Margolis DA, Smith KY, Vanveggel S, Spreen W. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 48-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet. 2021 Dec 19;396(10267):1994-2005. doi: 10.1016/S0140-6736(20)32666-0. Epub 2020 Dec 9. PMID 33308425
- [Result] Jaeger H, Overton ET, Richmond G, Rizzardini G, Andrade-Villanueva JF, Mngqibisa R, Hermida AO, Thalme A, Belonosova E, Ajana F, Benn PD, Wang Y, Hudson KJ, Espanol CM, Ford SL, Crauwels H, Margolis DA, Talarico CL, Smith KY, van Eygen V, Van Solingen-Ristea R, Vanveggel S, Spreen WR. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 96-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet HIV. 2021 Nov;8(11):e679-e689. doi: 10.1016/S2352-3018(21)00185-5. Epub 2021 Oct 11. PMID 34648734
- [Result] Orkin C, Oka S, Philibert P, Brinson C, Bassa A, Gusev D, Degen O, Garcia JG, Morell EB, Tan DHS, D'Amico R, Dorey D, Griffith S, Thiagarajah S, St Clair M, Van Solingen-Ristea R, Crauwels H, Ford SL, Patel P, Chounta V, Vanveggel S, Cutrell A, Van Eygen V, Vandermeulen K, Margolis DA, Smith KY, Spreen WR. Long-acting cabotegravir plus rilpivirine for treatment in adults with HIV-1 infection: 96-week results of the randomised, open-label, phase 3 FLAIR study. Lancet HIV. 2021 Apr;8(4):e185-e196. doi: 10.1016/S2352-3018(20)30340-4. PMID 33794181
- [Result] Cutrell AG, Schapiro JM, Perno CF, Kuritzkes DR, Quercia R, Patel P, Polli JW, Dorey D, Wang Y, Wu S, Van Eygen V, Crauwels H, Ford SL, Baker M, Talarico CL, Clair MS, Jeffrey J, White CT, Vanveggel S, Vandermeulen K, Margolis DA, Aboud M, Spreen WR, van Lunzen J. Exploring predictors of HIV-1 virologic failure to long-acting cabotegravir and rilpivirine: a multivariable analysis. AIDS. 2021 Jul 15;35(9):1333-1342. doi: 10.1097/QAD.0000000000002883. PMID 33730748
- [Result] Cooper V, Clatworthy J, Harding R, Whetham J; Emerge Consortium. Measuring quality of life among people living with HIV: a systematic review of reviews. Health Qual Life Outcomes. 2017 Nov 15;15(1):220. doi: 10.1186/s12955-017-0778-6. PMID 29141645
- [Result] Wu AW, Hanson KA, Harding G, Haider S, Tawadrous M, Khachatryan A, Pashos CL, Simpson KN. Responsiveness of the MOS-HIV and EQ-5D in HIV-infected adults receiving antiretroviral therapies. Health Qual Life Outcomes. 2013 Mar 12;11:42. doi: 10.1186/1477-7525-11-42. PMID 23497257
- [Result] Tatlock S, Arbuckle R, Sanchez R, Grant L, Khan I, Manvelian G, Spertus JA. Psychometric Evaluation of a Treatment Acceptance Measure for Use in Patients Receiving Treatment via Subcutaneous Injection. Value Health. 2017 Mar;20(3):430-440. doi: 10.1016/j.jval.2016.09.2410. Epub 2016 Dec 1. PMID 28292488
- [Result] Chounta V, Overton ET, Mills A, Swindells S, Benn PD, Vanveggel S, van Solingen-Ristea R, Wang Y, Hudson KJ, Shaefer MS, Margolis DA, Smith KY, Spreen WR. Patient-Reported Outcomes Through 1 Year of an HIV-1 Clinical Trial Evaluating Long-Acting Cabotegravir and Rilpivirine Administered Every 4 or 8 Weeks (ATLAS-2M). Patient. 2021 Nov;14(6):849-862. doi: 10.1007/s40271-021-00524-0. Epub 2021 May 31. PMID 34056699
- [Result] Swindells S, Lutz T, Van Zyl L, Porteiro N, Stoll M, Mitha E, Shon A, Benn P, Huang JO, Harrington CM, Hove K, Ford SL, Talarico CL, Chounta V, Crauwels H, Van Solingen-Ristea R, Vanveggel S, Margolis DA, Smith KY, Vandermeulen K, Spreen WR. Week 96 extension results of a Phase 3 study evaluating long-acting cabotegravir with rilpivirine for HIV-1 treatment. AIDS. 2022 Feb 1;36(2):185-194. doi: 10.1097/QAD.0000000000003025. PMID 34261093
- [Result] Karver TS, Pascual-Bernaldez M, Berni A, Hnoosh A, Castagna A, Messiaen P, Puerto MJG, Bloch M, Adachi E, Sinclair G, Felizarta F, Angel JB, Sutton K, Sutherland-Phillips D, D'Amico R, Kerrigan D. Factors Associated with Health Care Providers' Preference for Forgoing an Oral Lead-In Phase When Initiating Long-Acting Injectable Cabotegravir and Rilpivirine in the SOLAR Clinical Trial. AIDS Patient Care STDS. 2023 Jan;37(1):53-59. doi: 10.1089/apc.2022.0168. PMID 36626155
- [Result] Orkin C, Bernal Morell E, Tan DHS, Katner H, Stellbrink HJ, Belonosova E, DeMoor R, Griffith S, Thiagarajah S, Van Solingen-Ristea R, Ford SL, Crauwels H, Patel P, Cutrell A, Smith KY, Vandermeulen K, Birmingham E, St Clair M, Spreen WR, D'Amico R. Initiation of long-acting cabotegravir plus rilpivirine as direct-to-injection or with an oral lead-in in adults with HIV-1 infection: week 124 results of the open-label phase 3 FLAIR study. Lancet HIV. 2021 Nov;8(11):e668-e678. doi: 10.1016/S2352-3018(21)00184-3. Epub 2021 Oct 14. PMID 34656207
- See also: Panel on Treatment of HIV During Pregnancy and Prevention of Perinatal Transmission. Recommendations for Use of Antiretroviral Drugs in Transmission in the United States. — https://clinicalinfo.hiv.gov/en/guidelines/perinatal/whats-new
- See also: A Study to Evaluate Efficacy and Safety of Cabotegravir (CAB) Long Acting (LA) Plus (+) Rilpivirine (RPV) LA Versus BIKTARVY® (BIK) in Participants With Human Immunodeficiency Virus (HIV)-1 Who Are Virologically Suppressed — http://ClinicalTrials.gov
- See also: Information leaflet for professionals VOCABRIA prolonged-release injectable suspension 600 mg/3ml. — http://www.ispch.cl/wp-content/uploads/2021/10/F-26400.pdf
- See also: Use of cabotegravir and rilpivirine tablets to control the planned interruption of the injection dose every 2 months with cabotegravir long-acting plus rilpivirine. ViiV Healthcare — https://d201nm4szfwn7c.cloudfront.net/5f95dbd7-245e-4e65-9f36-1a99e28e5bba/1f05f316-0871-4693-843d-5a8da162e5d7/1f05f316-0871-4693-843d-5a8da162e5d7_viewable_rendition__v.pdf
- See also: HIGHLIGHTS OF PRESCRIBING INFORMATION — http://www.accessdata.fda.gov
- See also: Information leaflet for ptofessionals Vocabria prolonged-release injectable suspension 600 mg/3ml. updated — https://www.ispch.gob.cl/wp-content/uploads/2022/09/F_26400.pdf